CLINICAL TRIAL: NCT01565343
Title: Test-retest Reproducibility of 18F-AV-45 for Brain Imaging of Amyloid in Healthy Volunteers and Alzheimer's Disease Patients
Brief Title: A Study of 18F-AV-45 in Alzheimer's Disease (AD) and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A04
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer's Disease
Keywords: Amyloid imaging; Positron Emission Tomography; 18F-AV-45; florbetapir F 18; Diagnostic imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AD Subjects (Experimental): Two bolus IV injections followed by brain PET scan up to 4 weeks apart
  Interventions: Drug: florbetapir F 18
- AD Subjects: Slow vs. Fast Bolus (Experimental): Two bolus IV injections followed by a brain PET scan up to 4 weeks apart.
  The first injection given as a rapid bolus (< 5 second injection, with immediate flush). The second injection given as a slow bolus (approximately 20 to 30 second injection with a flush delayed by 10 seconds after dose administration).
  Interventions: Drug: florbetapir F 18
- Healthy controls (Experimental): Healthy male or female subjects; 35-55 years old. Two bolus IV injections followed by brain PET scan up to 4 weeks apart
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — IV injection, 370MBq (10mCi)
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
This study will test if two AV-45 PET scans up to 4 weeks apart in AD subjects and healthy volunteers provide the same results. The study will also test two different AV-45 injection methods in a small subgroup of enrolled AD subjects (slow vs. fast bolus group).

ELIGIBILITY:
Inclusion Criteria (AD group):

* Greater than 50 years of age
* Probable AD according to the National Institute of Neurological and Communication Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Mild/moderate dementia as evidenced by a Mini-Mental State Examination (MMSE) score ranging from 10 to 24, boundaries included, at screening
* History of cognitive decline gradual in onset and progressive over a period of at least 6 months

Inclusion Criteria (healthy volunteer group):

* 35 to 55 years of age, inclusive
* MMSE of 29 or greater

Exclusion Criteria (both groups):

* Neurodegenerative disorders other than AD, including, but not limited to Parkinson's disease, Pick's disease, fronto-temporal dementia, Huntington's chorea, Down syndrome, Creutzfeldt-Jacob disease, normal pressure hydrocephalus, and progressive supranuclear palsy
* Diagnosis of other dementing / neurodegenerative disease
* Diagnosis of mixed dementia
* Cognitive impairment resulting from trauma, hypoxic damage, vitamin deficiency, brain infection, brain cancer, endocrine disease, or mental retardation
* Clinically significant infarct or possible multi-infarct dementia as defined by the NINCDS criteria
* Evidence on screening MRI or other biomarker that suggests alternate etiology for cognitive deficit (for healthy controls, evidence suggesting the presence of AD pathology)
* Clinically significant psychiatric disease
* History of epilepsy or convulsions
* Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances
* Current clinically significant cardiovascular disease
* Received investigational medication within the last 30 days

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (4):
- United States (4):
  - Research Site, New Haven, Connecticut
  - Research Site, Hallandale, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, North East, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- AD Subjects: Male or female subjects > 50 years old; probable AD according to NINCDS-ADRDA criteria; MMSE 10-24
- AD Subjects: Slow vs. Fast Bolus Group: Same inclusion criteria as AD subjects. The first injection given as a rapid bolus (< 5 second injection, with immediate flush). The second injection given as a slow bolus (approximately 20 to 30 second injection with a flush delayed by 10 seconds after dose administration).
- Control Subjects: Healthy male or female subjects; 35-55 years old; no evidence of cognitive impairment; MMSE 29 or higher
Period: Overall Study
Arm/Group | AD Subjects | AD Subjects: Slow vs. Fast Bolus Group | Control Subjects
Started | 11 | 4 | 10
Completed | 10 | 4 | 10
Not Completed | 1 | 0 | 0
Not completed — Administrative decision/technical issues | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AD Subjects | AD Subjects: Slow vs. Fast Bolus Group | Control Subjects | Total
Number analyzed (Participants) | 11 | 4 | 10 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 69.7 (10.66) | 79.0 (3.56) | 44.4 (5.64) | 61.1 (16.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 4 | 16
  Male | 2 | 1 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 11 | 4 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Cortical to Cerebellum SUVR
Description: Standardized Uptake Value ratio (SUVR) is the ratio of tracer uptake in predefined cortical regions, relative to uptake in the whole cerebellum.
Time Frame: 50-70 min after injection
Population: Due to poor subject positioning that resulted in an incomplete brain image on the retest image day, accurate quantitative analysis for one healthy control was not possible, and the subject was excluded from the SUVR-based analyses.
Measure: Mean (Standard Deviation); unit: SUVR
Groups:
- AD Subjects: Male or female subjects > 50 years old; probable Alzheimer's Disease) AD according to National Institute of Neurological and Communication Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria; Mini-Mental State Examination (MMSE) 10-24
Arm/Group | AD Subjects | Control Subjects
Number analyzed (Participants) | 10 | 9
SUVR
  Test (50-70 min) | 1.416 (0.245) | 1.005 (0.055)
  Retest (50-70 min) | 1.407 (0.269) | 1.007 (0.061)
Statistical Analysis 1: Comparison: AD Subjects; Intra-class Correlation Coefficient (ICC) of AD subjects 50-70 min test vs. retest values; Test type: Superiority or Other; ICC; ICC = 0.9893
Statistical Analysis 2: Comparison: Control Subjects; Intra-class Correlation Coefficient of Control subjects 50-70 min test vs. retest values; Test type: Superiority or Other; ICC; ICC = 0.9574
Statistical Analysis 3: Comparison: AD Subjects; Intra-subject variability (% difference) of AD subjects 50-70 min test vs. retest values; Test type: Superiority or Other; Mean % difference = 2.35, Standard Deviation 1.413
Statistical Analysis 4: Comparison: Control Subjects; Intra-subject variability (% difference) of control subjects 50-70 min test vs. retest values; Test type: Superiority or Other; Mean % difference = 1.49, Standard Deviation 0.839

ADVERSE EVENTS:
Time Frame: AEs reported within 7 days of injection. SAEs reported within 30 days of injection.
Arm/Group | AD Subjects | AD Subjects: Slow vs. Fast Bolus Group | Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/4 | 0/10
Other Adverse Events (participants affected / at risk) | 1/11 | 0/4 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AD Subjects (N=11) | AD Subjects: Slow vs. Fast Bolus Group (N=4) | Control Subjects (N=10)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days